CLINICAL TRIAL: NCT00495079
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Weekly Doses of Marqibo® (Vincristine Sulfate Liposomes Injection) in Adult Patients With Philadelphia Chromosome-negative Acute Lymphoblastic Leukemia (ALL) in Second Relapse or Adult Patients With Philadelphia Chromosome-negative ALL Who Failed Two Treatment Lines of Anti-leukemia Chemotherapy
Brief Title: Safety and Efficacy of Marqibo in Relapsed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBS407
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
Keywords: acute; lymphoblastic; lymphocytic; leukemia; leukaemia; lukemia; leukimia; ALL; Marqibo; Hana Biosciences; vincristine; liposomal; liposome; optisome; hematology; malignancy; hematological; relapsed; anti-leukemia; adult; chemotherapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Neoplasms; Recurrence | interventions — Vincristine

ARMS (1):
- Marqibo (Experimental): Eligible subjects received study drug at 2.25 mg/m^2 intravenously via peripheral or central venous access over 60 minutes (± 10 minutes).
  Interventions: Drug: Marqibo® (vincristine sulfate liposomes injection)

INTERVENTIONS:
Drug: Marqibo® (vincristine sulfate liposomes injection) — Dosing was done every 7 days (± 3 days) on Days 1, 8, 15, and 22 with no less than 4 days between dosing days. Dose calculations were based on body surface area using the subject's height (from Screening) and actual weight for each course.
  Other Names: VSLI, Vincristine Sulfate Liposomes Injection

SUMMARY:
This was a Phase 2, international, multicenter, open-label, single-arm trial evaluating Marqibo (VSLI) in adult subjects with: 1) Ph- ALL or lymphoblastic lymphoma in second or greater relapse; or 2) Ph- ALL or lymphoblastic lymphoma who failed 2 or greater treatment lines of anti-leukemia chemotherapy. The original enrollment target for this study was approximately 56 subjects. Per a protocol amendment, enrollment was increased from 56 to 65.

The primary objective of this study was to evaluate:

- The efficacy of the study treatment as determined by the rate of CR plus CR with incomplete blood count recovery (CRi) in adult subjects with Philadelphia chromosome-negative (Ph-) ALL in second relapse or adult subjects with (Ph-) ALL who failed 2 treatment lines of anti-leukemia chemotherapy. Subjects must have achieved a CR to at least 1 prior anti-leukemia therapy as defined by a leukemia-free interval of ≥ 90 days.

DETAILED DESCRIPTION:
The secondary objectives of this study were to evaluate:

* Duration of CR plus CRi
* Overall survival
* Safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Had Ph- ALL or lymphoblastic lymphoma and was in second relapse, or had failed 2 treatment lines of anti-leukemia chemotherapy.
* Had histologically or cytologically proven ALL and ≥ 10% bone marrow blasts. If < 10% bone marrow blasts, subject must have had histologically or cytologically proven ALL and evaluable extramedullary disease. Sponsor approval was obtained prior to enrolling subjects who had < 10% bone marrow blasts with evaluable extramedullary disease.
* Had achieved a CR to at least 1 prior anti-leukemia therapy as defined by a leukemia-free interval of ≥ 90 days.
* For subjects with a prior history of stem cell transplantation, had ≤ Grade 1 active skin graft-versus-host disease (GVHD). No active gastrointestinal or liver graft-versus-host disease.
* Had an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 3.
* Had normal renal and liver function as defined below within 14 days, inclusive, prior to first dose of VSLI, unless the abnormality was considered attributable to leukemia:
* Total bilirubin ≤ 2.0 × institutional upper limit of normal, unless the subject had a known diagnosis of Gilbert's disease. If a subject had Gilbert's disease, he/she could have participated in this study, however must have been monitored closely during the study.
* Aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 3 × institutional upper limit of normal.
* Serum creatinine ≤ 2.0 g/dL or calculated estimated creatinine clearance ≥ 50 mL/minute/1.73 m2 based on Cockcroft and Gault formula, unless renal dysfunction was considered due to hematologic malignancy.
* Had never received prior VSLI treatment.
* For women of childbearing potential, had a negative serum or urine pregnancy test within 14 days prior to enrollment.
* If female, the subject was postmenopausal, surgically sterilized, or willing to use acceptable methods of birth control (e.g., hormonal contraceptive, intra-uterine device, diaphragm with spermicide, and condom with spermicide or abstinence) from the Screening visit through 30 days after the last dose of VSLI.
* If male, the subject agreed to use an acceptable barrier method for contraception from the Screening visit through 30 days after the last dose of VSLI.
* Before enrollment, the subject was capable of understanding and complying with parameters as outlined in the protocol and able to sign a written informed consent according to ICH/GCP and national/local regulations.

Exclusion Criteria:

* Had Burkitt's lymphoma or Burkitt's leukemia.
* Had a history of Philadelphia chromosome-positive (Ph+) ALL and/or BCR/ABL rearrangements documented by fluorescent in situ hybridization or polymerase chain reaction.
* Had a history of Philadelphia chromosome-positive (Ph+) ALL and/or BCR/ABL rearrangements documented by fluorescent in situ hybridization or polymerase chain reaction.
* Had active CNS disease. History of treated CNS disease was allowable. The CNS disease must have resolved in order for the subject to be eligible.
* Was eligible for stem cell transplantation. This implied that a suitable donor was readily available, the subject was willing to undergo stem cell transplantation, and the Investigator believed this was a better treatment option than VSLI. This was at the Investigator's discretion.
* Was treated with any investigational agents or chemotherapy agents in the last 21 days before the first dose of VSLI, unless full recovery from side effects had occurred or the subject had rapidly progressing disease judged to be life threatening by the Investigator.
* Was receiving any other standard or investigational treatment for the subject's leukemia.
* Intrathecal chemotherapy for CNS prophylaxis was allowable.
* The use of hydroxyurea (Hydrea®) to control leukocytosis was allowable but must have been tapered off by Day 14 of Course 1. From Day 15 of Course 1 on through the end of study participation, hydroxyurea (Hydrea®) was not allowed.
* Systemic corticosteroids must have been tapered off, preferably before the start of study treatment, but no later than by Day 5 of Course 1. From Day 6 of Course 1 on through the end of study participation, systemic corticosteroids were not allowed.
* Had persistent chronic clinically significant toxicities from prior chemotherapy ≥ Grade 2 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 3.0).
* Had persistent ≥ Grade 2 active neuropathy (NCI CTCAE v3.0).
* Had a history of persistent ≥ Grade 2 active neurologic disorders unrelated to chemotherapy (including demyelinating form of Charcot-Marie-Tooth syndrome, acquired demyelinating disorders, or other demyelinating condition).
* Had a history of allergic reactions or sensitivity attributed to compounds of similar chemical or biologic composition to vincristine or components of study drug.
* Was female who was pregnant or breast-feeding.
* Had active serious infection not controlled by oral or intravenous antibiotics or antifungals.
* Had human immunodeficiency virus positive status.
* Had any medical condition which in the opinion of the investigator placed the subject at an unacceptably high risk for toxicities.
* Had any condition or circumstance which in the opinion of the investigator would significantly interfere with the subject's protocol compliance and put the subject at increased risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-05; Primary Completion 2010-08-08 (Actual); Study Completion 2010-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan O'Brien, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (33):
- United States (18):
  - USC - Norris Cancer Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - University of California Medical Center, San Francisco, California
  - Stanford Hospitals and Clinics, Stanford, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Loyola University Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Univesity of Iowa - Hospitals and Clinica, Iowa City, Iowa
  - Henry Ford Health System, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Medical College, Valhalla, New York
  - Western Pennsylvania Allegheny Health System, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Germany (9):
  - Dresden University Hospital, Dresden
  - University of Essen, Essen
  - J.W. Goethe University, Frankfurt
  - University of Leipzig, Leipzig
  - University of Muenster, Münster
  - University of Rostock, Rostock
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Robert Bosch Hospital, Stuttgart
  - University of Ulm, Ulm
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center - Ein Karem, Jerusalem
  - Rabin Medical Center Campus, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Derriford Hospital, Plymouth, United Kingdom

REFERENCES:
- [Derived] Schiller GJ, Damon LE, Coutre SE, Hsu P, Bhat G, Douer D. High-Dose Vincristine Sulfate Liposome Injection, for Advanced, Relapsed, or Refractory Philadelphia Chromosome-Negative Acute Lymphoblastic Leukemia in an Adolescent and Young Adult Subgroup of a Phase 2 Clinical Trial. J Adolesc Young Adult Oncol. 2018 Oct;7(5):546-552. doi: 10.1089/jayao.2018.0041. Epub 2018 Sep 21. PMID 30239252
- [Derived] Silverman JA, Reynolds L, Deitcher SR. Pharmacokinetics and pharmacodynamics of vincristine sulfate liposome injection (VSLI) in adults with acute lymphoblastic leukemia. J Clin Pharmacol. 2013 Nov;53(11):1139-45. doi: 10.1002/jcph.155. Epub 2013 Aug 17. PMID 23907766
- [Derived] O'Brien S, Schiller G, Lister J, Damon L, Goldberg S, Aulitzky W, Ben-Yehuda D, Stock W, Coutre S, Douer D, Heffner LT, Larson M, Seiter K, Smith S, Assouline S, Kuriakose P, Maness L, Nagler A, Rowe J, Schaich M, Shpilberg O, Yee K, Schmieder G, Silverman JA, Thomas D, Deitcher SR, Kantarjian H. High-dose vincristine sulfate liposome injection for advanced, relapsed, and refractory adult Philadelphia chromosome-negative acute lymphoblastic leukemia. J Clin Oncol. 2013 Feb 20;31(6):676-83. doi: 10.1200/JCO.2012.46.2309. Epub 2012 Nov 19. PMID 23169518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled and treated at 22 sites in United States, Canada, Germany, Israel and United Kingdom. The first subject was infused on August 2, 2007. The last subject completed study on August 8, 2010.
Pre-assignment Details: 2.25 mg/m^2 Marqibo administered intravenously via peripheral or central venous access over 60 minutes (+-10 minutes)
Groups:
- Marqibo: Eligible subjects received study drug at 2.25 mg/m2 intravenously via peripheral or central venous access over 60 minutes (± 10 minutes).
Period: Overall Study
Arm/Group | Marqibo
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Marqibo
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 59
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (16.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 53
  Canada | 2
  Israel | 6
  Germany | 4

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Plus Complete Remission Without Full Platelet Recovery (CR + CRi)
Description: CR is defined as no evidence of ALL: ANC>or=1x10^9/L or platelet count>100x10^9/L, absence of leukemia blast cells in blood and marrow (<5% blasts), resolution of all sites of extramedullary disease (EMD). CR with incomplete blood count recovery (CRi): As per CR but platelet count< 100x10^9/L or ANC< 1x10^9/L. Partial remission(PR):CR with>5-25% abnormal cells in the marrow or 50% decrease in bone marrow blasts. Reduction in EMD by at least 50%. Hematologic Improvement. Bone marrow blast(BMB) response: BMB<5% in the absence of HI. Stable disease(SD):No significant hematological and extramedullary change from baseline.
Time Frame: Response assessment performed at the end of each 28 day course.
Population: Subjects who had CR plus CRi by the PI and the IRRC assessments using the International Working Group Criteria. The Intent-to-Treat Analysis, n=65, minimum 1 dose. The IRRC, n=53, 1 dose, assess response as determined by the IRRC. Analyses, a Simon's 2-stage minimax design where the type I error alpha was set at 0.10 and the power was 80%.
Measure: Number; unit: participants
Arm/Group | Marqibo
Number analyzed (Participants) | 65
participants | 13 [11.1 to 31.8]

2. Secondary Outcome: Duration of CR + CRi
Description: Duration of response for those subjects who achieved CR or CRi
Time Frame: CR + CRi duration was calculated from the date the subject first met the definition of CR or CRi until the date of relapse
Population: Based on the first date of CR or CRi to the date of the last available histologic assessment of the same response (n=8)
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Marqibo: Duration of response derived using the IRRC determined response dates for subjects who achieved CR or CRi (n=8). The K-M product limit method was used to estimate the median event time.
  Eligible subjects received Marqibo at 2.25mg^m2 intravenously via peripheral or central venous access over 60 minutes (+- 10 minutes)every 7 days (+/- 3 days)
Arm/Group | Marqibo
Number analyzed (Participants) | 8
days | 28 [7 to 36]

3. Secondary Outcome: Overall Survival
Description: Time, in days, from informed consent date until the date of death or date of last contact
Time Frame: unlimited
Population: Based on the first date of CR or CRi to date of documented relapse, death, or subsequent chemotherapies including hematopoietic stem cell transplant (HSCT)(n=10)
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Marqibo: The population analyzed included all subjects who received at least one dose of Marqibo. Subjects who did not die had their survival times censored on the date of last contact. The K-M method was used to estimate the distribution of overall survival.
  Eligible subjects received study drug at 2.25 mg/m2 intravenously via peripheral or central venous access over 60 minutes (± 10 minutes)every 7 days (+/- 3 days)
Arm/Group | Marqibo
Number analyzed (Participants) | 10
days | 56 [9 to 65]

4. Primary Outcome: Clinical Response Assessment Per Independent Response Review Committee (IRRC) Evaluation
Description: Number of subjects who achieved Complete Remission (CR)as assessed by the IRRC. CR is defined as no evidence of ALL. ANC>=1X10^9/L or Platelet count>=100x10^9/L, absence of blasts in blood and morrow (<5%), resolution of all sites of extramedullary disease (EMD). CR with incomplete blood count recovery(CRi)is defined as per CR but platelet count <100x10^9/L or ANC<1x10^9/L.
Time Frame: Response assessment at the end of each 28 days course
Population: The IRRC evaluable population included all subjects who received at least 1 dose of study drug and who has reviewable data to assess and determine response or lack of response as determined by the IRRC.
Measure: Number; unit: participants
Groups:
- Marqibo: Proportion if subjects who achieved CR+CRi as determined by the IRRC using the International Working Group (IWG)Criteria. The IRRC Evaluable analysis set(n=53) included subjects who received at least 1 dose of study drug and reviewable data.
  Eligible subjects received Marqibo at 2.25mg^m2 intravenously via peripheral or central venous access over 60 minutes (+/-10 minutes) every 7 days (+/-3days)
Arm/Group | Marqibo
Number analyzed (Participants) | 53
participants | 11 [10.8 to 34.1]

ADVERSE EVENTS:
Time Frame: From date of first dose of study drug until 30 days after last Marqibo dose (+ 5 days)
Arm/Group | Marqibo
Serious Adverse Events (participants affected / at risk) | 21/65
Other Adverse Events (participants affected / at risk) | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marqibo (N=65)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (12)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Neuropathy, peripheral (Nervous system disorders) | 4 (4)
Facial palsy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropath (Nervous system disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Cholecystitis, chronic (Hepatobiliary disorders) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Venoocclusive disease (Vascular disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) — 1
Sepsis (Infections and infestations) | 2 (2)
Septic Shock (Infections and infestations) | 2 (2)
Acute Sinusitis (Infections and infestations) | 1 (1)
Bronchiectasis (Infections and infestations) | 1 (1)
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Entrocococcal Bacteraemia (Infections and infestations) | 1 (1)
Escherichia Sepsis (Infections and infestations) | 1 (1)
Klebsiella Sepsis (Infections and infestations) | 1 (1)
Neutropenic Sepsis (Infections and infestations) | 1 (1)
Parainfluenzae Virus Infection (Infections and infestations) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Acute Lymphocytic Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9)
Acute Lymphocytic Leukaemia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia Infiltration Brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Heamorrhage Intracranial (Nervous system disorders) | 1 (1)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1)
Gait Disturbance (General disorders) | 1 (1)
Multi-Organ Failure (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 3 (3)
Cardio-Respiratory Arrest (Cardiac disorders) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Mental Status Changes (Psychiatric disorders) | 2 (2)
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Csf Bacteria Identified (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marqibo (N=65)
Nausea (Gastrointestinal disorders) | 35 (35)
Constipation (Gastrointestinal disorders) | 34 (34)
Diarrhoea (Gastrointestinal disorders) | 22 (22)
Vomiting (Gastrointestinal disorders) | 17 (17)
Abdominal pain (Gastrointestinal disorders) | 13 (13)
Stomatitis (Gastrointestinal disorders) | 9 (9)
Abdominal distension (Gastrointestinal disorders) | 7 (7)
Gingival bleeding (Gastrointestinal disorders) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 4 (4)
Pyrexia (General disorders) | 25 (25)
Fatigue (General disorders) | 19 (19)
Asthenia (General disorders) | 15 (15)
Pain (General disorders) | 15 (15)
Oedema, peripheral (General disorders) | 10 (10)
Chills (General disorders) | 8 (8)
Chest pain (General disorders) | 7 (7)
Neuropathy, peripheral (Nervous system disorders) | 20 (20)
Headache (Nervous system disorders) | 17 (17)
Hypoaesthesia (Nervous system disorders) | 16 (16)
Paraesthesia (Nervous system disorders) | 14 (14)
Dizziness (Nervous system disorders) | 10 (10)
Areflexia (Nervous system disorders) | 6 (6)
Hyporeflexia (Nervous system disorders) | 5 (5)
Cranial neuropathy (Nervous system disorders) | 4 (4)
Facial neuralgia (Nervous system disorders) | 4 (4)
Neuralgia (Nervous system disorders) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 24 (24)
Anaemia (Blood and lymphatic system disorders) | 17 (17)
Neutropenia (Blood and lymphatic system disorders) | 15 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (15)
Leukopenia (Blood and lymphatic system disorders) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 24 (24)
Hypokalaemia (Metabolism and nutrition disorders) | 17 (17)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (9)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 5 (5)
Cachexia (Metabolism and nutrition disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Weight decreased (Investigations) | 10 (10)
Alanine aminotransferase increased (Investigations) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 7 (7)
Blood lactate dehydrogenase increased (Investigations) | 7 (7)
Blood alkaline phosphatase increased (Investigations) | 4 (4)
Insomnia (Psychiatric disorders) | 16 (16)
Confusional state (Psychiatric disorders) | 10 (10)
Anxiety (Psychiatric disorders) | 6 (6)
Depression (Psychiatric disorders) | 5 (5)
Agitation (Psychiatric disorders) | 4 (4)
Pneumonia (Infections and infestations) | 9 (9)
Oral candidiasis (Infections and infestations) | 4 (4)
Septic shock (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 8 (8)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4)
Hypertension (Vascular disorders) | 11 (11)
Hypotension (Vascular disorders) | 10 (10)
Orthostatic hypotension (Vascular disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 11 (11)
Urinary incontinence (Renal and urinary disorders) | 4 (4)
Acute lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less